CLINICAL TRIAL: NCT03030378
Title: A Phase 1 Study of Pembrolizumab (MK-3475) in Combination With Recombinant Interleukin-12 in Patients With Solid Tumors
Brief Title: Pembrolizumab and Recombinant Interleukin-12 in Treating Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00091; NCI-2017-00091 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCC 17-003; 10061 (Other: UPMC Hillman Cancer Center LAO); 10061 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-25 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Interleukin-12; Interleukin-12 Subunit p35; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (recombinant interleukin-12, pembrolizumab) (Experimental): Patients receive recombinant interleukin-12 SC on days 2, 5, 9, and 12 and pembrolizumab IV over 30 minutes on day 8 of cycle 1 and day 1 of subsequent cycles. Treatment continues for 28 days for cycle 1 and repeats every 21 days for subsequent cycles for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patient then receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 8 additional cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT, PET, and MRI, as well as collection of blood during screening, on study, and during follow-up. Patients also undergo a tumor biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Edodekin alfa; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo a tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Edodekin alfa — Given SC
  Other Names: Cytotoxic Lymphocyte Maturation Factor; IL-12; Interleukin 12; Interleukin-12; Natural Killer Cell Stimulatory Factor; NM-IL-12; Recombinant human interleukin-12 (IL-12) cytokine; Ro 24-7472
Procedure: Magnetic Resonance Imaging — Undergo a MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo a PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial studies the side effects and best dose of pembrolizumab and recombinant interleukin-12 in treating patients with solid tumors. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Recombinant interleukin-12 may kill tumor cells by blocking blood flow to the tumor and by stimulating white blood cells to kill tumor cells. Giving pembrolizumab and recombinant interleukin-12 may work better than giving pembrolizumab alone in treating patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Establish the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of edodekin alfa (recombinant human interleukin [rhIL]-12) in combination with pembrolizumab (MK-3475).

SECONDARY OBJECTIVES:

I. Evaluate the safety of the regimen by continuously monitoring adverse events that will be documented utilizing Common Terminology Criteria for Adverse Events (CTCAE) version (v).5.0.

II. Evaluate the overall response rate (Response Evaluation Criteria in Solid Tumors [RECIST] v.1.1) and the progression free survival of patients enrolled on the study.

III. Measure CD8+ T cell infiltration by immunohistochemistry in tumor biopsies obtained pre-treatment, after one week of rhIL-12 and after 2 cycles of pembrolizumab (MK-3475) in combination with rhIL-12.

EXPLORATORY OBJECTIVE:

I. Conduct exploratory translational laboratory correlative studies utilizing banked biospecimens (tumor, blood, and stool) obtained pre-treatment and during therapy.

OUTLINE: This is a dose-escalation study of recombinant interleukin-12.

Patients receive recombinant interleukin-12 subcutaneously (SC) on days 2, 5, 9, and 12 and pembrolizumab intravenously (IV) over 30 minutes on day 8 of cycle 1 and day 1 of subsequent cycles. Treatment continues for 28 days for cycle 1 and repeats every 21 days for subsequent cycles for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patient then receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 8 additional cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a computed tomography (CT), positron emission tomography (PET), and/or magnetic resonance imaging (MRI), as well as collection of blood during screening, on study, and during follow-up. Patients also undergo a tumor biopsy during screening and on study.

After completion of study treatment, patients are followed up every 12 weeks for 2 year and then every 24 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable
* Eligibility is restricted to patients who have tumors for which there is a Food and Drug Administration (FDA)-approved indication for anti-PD-(L)1 therapy. Patients must have received and have progressed past anti-PD(L)1 singly or in combination. There is no restriction on the number of prior lines of therapy. Anti-PD-(L)1 therapy need not be the most recent therapy received

  * NOTE: Prior to slot reservation, sites must provide the following information to ETCTN10061@upmc.edu for study chair review: histology, nature of prior therapy (therapies) and indication for prior PD-(L)1 therapy
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of pembrolizumab (MK-3475) in combination with rhIL-12 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 2,000/mcL (within 28 days of treatment initiation)
* Absolute neutrophil count >= 1,500/mcL (within 28 days of treatment initiation)
* Platelets >= 100,000/mcL (within 28 days of treatment initiation)
* Hemoglobin >= 9 g/dL OR >= 5.6 mmol/L (within 28 days of treatment initiation)
* Serum total bilirubin =< upper limit of normal (ULN) OR direct bilirubin =< ULN for patients with total bilirubin levels > ULN; (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL) (within 28 days of treatment initiation)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 x institutional ULN (within 28 days of treatment initiation)
* Serum creatinine =< 1.5 x ULN OR measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (within 28 days of treatment initiation)

  * Creatinine clearance should be calculated per institutional standard
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as (PT) or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 28 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as prothrombin time (PT) or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 28 days of treatment initiation)
* Willingness to undergo tumor biopsies at three timepoints: (1) pre-treatment; (2) after one week of rhIL12; and (3) after 2 cycles of pembrolizumab (MK-3475)-interleukin (IL) 12 (i.e., approximately 7 weeks from the first dose of rhIL-12)

  * At each timepoint, a core biopsy is preferable (although in suitable patients, punch biopsy may be substituted)

    * Cytopathologist should be present to ensure adequacy of tumor biopsy sample
    * At least 4 16 gauge (G) core biopsies are to be obtained and triaged
  * Pre-treatment biopsy can be substituted with an archival tissue sample if the sample is

    * Adequate (capable of providing at least 20 unstained slides); and
    * Recent (within 8 weeks of study entry); and
    * Patient has not had any intervening therapy
* Patients must have measurable disease based on RECIST 1.1
* The effects of pembrolizumab (MK-3475) and/or rIL-12 on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

  * Female patients of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
  * Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of pembrolizumab (MK-3475) and/or rhIL-12 administration
* Ability to understand and the willingness to sign a written informed consent document
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * They must have an undetectable viral load
  * They must have a CD4 count of greater than 250 cells/mcL
  * They must not be receiving prophylactic therapy for an opportunistic infection

Exclusion Criteria:

* Patients with a secondary active hematological malignancy including but not limited to chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), Hodgkins lymphoma, non-Hodgkins lymphoma (NHL)

  * NOTE: Patients with a history of hematological malignancy that was previously treated and resolved may be enrolled if otherwise meeting inclusion/exclusion (I/E) criteria
* Patients with a prior history of autoimmune cytopenias of any etiology including hemolytic anemia, (AIHA), idiopathic thrombocytopenia purpura (ITP), and/or other cytopenia are excluded

  * NOTE: This exclusion is regardless of whether or not this cytopenia(s) required prior therapy
* Patients who have had chemotherapy, targeted small molecule therapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first dose of trial treatment, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

  * Note: Patients with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients who are currently participating in or have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of trial treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier; non-clinically significant adverse events may be considered as an exception after discussion with and approval by the principal investigator
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Patients with known active and untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with primary brain tumors or carcinomatous meningitis should also be excluded
* Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not requiring steroids for at least 7 days prior to trial treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab (MK-3475) and/or rhIL-12 or other agents used in study
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patients on any systemic corticosteroid therapy within one week before the planned date for first dose on study would not be eligible; exception: patients on physiologic replacement doses of corticosteroids are permitted
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment; pregnant women are excluded from this study because pembrolizumab (MK-3475) is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab (MK-3475), breastfeeding should be discontinued if the mother is treated with pembrolizumab (MK-3475); these potential risks may also apply to other agents used in this study; pembrolizumab (MK-3475) may have adverse effects on a fetus in utero; furthermore, it is not known if pembrolizumab (MK-3475) has transient adverse effects on the composition of sperm
* Men and non-pregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive; highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is >= 45 years of age and has not had menses for greater than 2 years will be considered postmenopausal), or 3) not heterosexually active for the duration of the study; the two birth control methods can be barrier method or a barrier method plus a hormonal method to prevent pregnancy; patients should start using birth control from study visit 1 throughout the study period up to 120 days after the last dose of study therapy; the following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide; appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents)

  * Patients should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study; in order to participate in the study they must adhere to the contraception requirement (described above) for the duration of the study and during the follow-up period; if there is any question that a patient will not reliably comply with the requirements for contraception, that patient should not be entered into the study
  * Pregnancy: If a patient inadvertently becomes pregnant while on treatment with pembrolizumab (MK-3475), the patient will immediately be removed from the study; the site will contact the patient at least monthly and document the patient's status until the pregnancy has been completed or terminated; the outcome of the pregnancy will be reported without delay and within 24 hours if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn); the study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn; if a male patient impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported and followed
  * It is unknown whether pembrolizumab (MK-3475) is excreted in human milk; since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, patients who are breast-feeding are not eligible for enrollment
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 5 years
Recommended phase 2 dose | Up to 5 years

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose
  Adverse events will be tabulated by Common Terminology Criteria for Adverse Events (CTCAE) grade, CTCAE category, relatedness to treatment and dose level.
Progression free survival | From start of treatment to time of progression or death, whichever comes, first assessed up to 5 years
  The product-limit (Kaplan-Meier) progression-free survival function, with a 95% confidence region, will be determined for all patients and for patients treated at the MTD.
Overall response rate | From start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started), assessed up to 5 years
  Will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1. The proportion of patients experiencing confirmed overall (complete or partial) response will be calculated, as will a 95% exact (Klopper-Pearson) binomial confidence interval for all patients, and patients treated at the MTD (a confirmed clinical tumor response is defined to be either a complete response or partial response noted as the objective status on 2 consecutive evaluations at least >= 4 weeks apart.).
CD8+ T cell infiltration | Up to 2 cycles of treatment
  Will be assessed by immunohistochemistry. Will be compared to pre-treatment biopsy specimens by the Wilcoxon signed-rank test.

OTHER OUTCOMES:
Biomarker analysis | Up to 5 years
  Will conduct exploratory translational laboratory correlative studies utilizing banked biospecimens (tumor, blood and stool) obtained at baseline and during therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (27):
- United States (27):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided